CLINICAL TRIAL: NCT04062201
Title: An Open Label, Randomized Controlled Trial to Establish the Efficacy and Safety of a Study Strategy Consisting of 6 Months of Bedaquiline (BDQ), Delamanid (DLM), and Linezolid (LNZ), With Levofloxacin (LVX) and Clofazimine (CFZ) Compared to the Current South African Standard of Care (Control Strategy) for 9 Months for the Treatment of Rifampicin Resistant Tuberculosis (RR-TB)
Brief Title: Building Evidence for Advancing New Treatment for Rifampicin Resistant Tuberculosis (RR-TB) Comparing a Short Course of Treatment (Containing Bedaquiline, Delamanid and Linezolid) With the Current South African Standard of Care
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wits Health Consortium (Pty) Ltd (Other)
Collaborators: Regents of the University of California (Other); University of Cape Town (Other); Perinatal HIV Research Unit of the University of the Witswatersrand (Other)
Responsible Party: Principal Investigator, Francesca Conradie, Deputy Director, Wits Health Consortium (Pty) Ltd
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BEAT Tuberculosis; 72067418CA00006 (Other Grant/Funding Number: USAID)
Record Dates: First submitted 2019-08-06; First posted 2019-08-20 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Tuberculosis; Pre-XDR-TB; Extensively Drug-Resistant Tuberculosis; Multi Drug Resistant Tuberculosis; Rifampicin Resistant Tuberculosis
Keywords: Tuberculosis; Drug-resistant Tuberculosis; Randomized Controlled Trial; Rifampicin Resistant Tuberculosis; Multi Drug Resistant Tuberculosis; Extensively Drug-Resistant Tuberculosis; Pre-XDR-TB (fluoroquinolone resistant); Open label; South Africa
MeSH Terms: conditions — Tuberculosis; Extensively Drug-Resistant Tuberculosis; Tuberculosis, Multidrug-Resistant | interventions — bedaquiline; Linezolid; OPC-67683; Dosage Forms; Clofazimine; Levofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Strategy (Experimental)
  Interventions: Drug: Bedaquiline Oral Tablet; Drug: Linezolid Oral Tablet; Drug: Delamanid in Oral Dosage Form; Drug: Clofazimine Oral Product; Drug: Levofloxacin Oral Tablet
- Control Strategy (Active Comparator)
  Interventions: Drug: Bedaquiline Oral Tablet; Drug: Isoniazid Oral Product; Drug: Ethambutol Oral Product; Drug: Pyrazinamide Oral Product; Drug: Linezolid Oral Tablet; Drug: Clofazimine Oral Product; Drug: Levofloxacin Oral Tablet

INTERVENTIONS:
Drug: Bedaquiline Oral Tablet — Weight Group 16 - 29.9kg: 200mg daily for two weeks; followed by 100mg three times weekly for weeks 3 - 24 Weight Group: 30 - >50kg: 400mg once daily for 14 days followed by 200mg three times weekly for weeks 3 - 24
  Other Names: Sirturo
Drug: Linezolid Oral Tablet — Weight Group 16 - 23kg: 180 - 210mg (crush 1 tab and mix in 10ml water, administer 3-3.5ml. Discard rest) Weight Group 23.1 - 29.9kg: 300mg daily Weight Group 30 - 33.9kg: 450mg daily Weight Group 34 - >50kg: 600mg daily
  Other Names: Zyvox
  Arms: Study Strategy
Drug: Delamanid in Oral Dosage Form — Weight Group 16 - 23kg: 25mg twice daily for 24 weeks Weight Group 23.1 - 33.9kg: 50mg twice daily for 24 weeks Weight Group 34 - >50kg: 100mg twice daily for 8 weeks followed by 200 mg daily for 16 weeks
  Other Names: Deltyba
  Arms: Study Strategy
Drug: Clofazimine Oral Product — Weight Group 16 - 23kg: 100mg three times a week or 50mg daily Weight Group 23.1 - >50kg: 100mg daily
  Other Names: Lamprene
  Arms: Study Strategy
Drug: Levofloxacin Oral Tablet — Weight Group 16 - 23kg: 375 - 500mg daily Weight Group 23.1 - 33.9kg: 500mg once daily Weight Group 34 - 50kg: 750mg daily Weight Group >50kg:1000mg daily
  Arms: Study Strategy
Drug: Isoniazid Oral Product — Weight Group 16 - 23kg: 300mg daily Weight Group 23.1 - 50kg: 400mg daily Weight Group >50kg: 600mg daily
  Other Names: INH
  Arms: Control Strategy
Drug: Ethambutol Oral Product — Weight Group 16 - 23kg: 400mg daily Weight Group 23.1 - 29.9kg: 600mg daily Weight Group 30 - 50kg: 800mg daily Weight Group >50kg: 1200mg daily
  Arms: Control Strategy
Drug: Pyrazinamide Oral Product — Weight Group 16 - 23kg: 750mg daily Weight Group 23.1 - 29.9kg: 1000mg daily Weight Group 30 - 33.9kg: 1250mg daily Weight Group 34 - 50kg: 1500mg daily Weight Group >50kg: 2000mg daily
  Arms: Control Strategy
Drug: Linezolid Oral Tablet — Weight Group 16 - 23kg: 180 - 210mg (crush 1 tab and mix in 10ml water, administer 3-3.5ml. Discard rest) Weight Group 23.1 - 29.9kg: 300mg daily Weight Group 30 - 33.9kg: 450mg daily Weight Group 34 - >50kg: 600mg daily
  Other Names: Zyvox
  Arms: Control Strategy
Drug: Clofazimine Oral Product — Weight Group 16 - 23kg: 100mg three times a week or 50mg daily Weight Group 23.1 - >50kg: 100mg daily
  Other Names: Lamprene
  Arms: Control Strategy
Drug: Levofloxacin Oral Tablet — Weight Group 16 - 23kg: 375 - 500mg daily Weight Group 23.1 - 33.9kg: 500mg once daily Weight Group 34 - 50kg: 750mg daily Weight Group >50kg:1000mg daily
  Arms: Control Strategy

SUMMARY:
BEAT Tuberculosis is a phase 3, open label, multi-centre, randomized controlled trial. The purpose of this trial is to compare the efficacy and safety of a Study Strategy consisting of 6 months of bedaquiline (BDQ), delamanid (DLM), and linezolid (LNZ), with levofloxacin (LVX) and clofazimine (CFZ) compared to the current South African Standard of Care (Control Strategy) for 9 months for the treatment of rifampicin resistant (RR-TB) Tuberculosis.

DETAILED DESCRIPTION:
In 2016, the World Health Organization (WHO) issued guidelines for the use of a shorter treatment regimen (STR) for eligible patients with RR and multidrug-resistant tuberculosis (MDR-TB) which was adopted by the South African National Tuberculosis Program (SANTP) in 2017. The WHO then released guidelines in September 2018 regrouping the medicines for the treatment of MDR/RR-TB into three categories and ranking them based on the latest evidence about the balance of effectiveness to safety. BDQ, LNZ and fluoroquinolones were moved to Category A and should be included in all regimens as core drugs. CFZ and terizidone as Category B drugs, should be added to all regimens.

The current short injectable-free treatment regimen for RR-TB in South Africa is based on these WHO recommendations. This South African standard of care, referred to as the Control Strategy, is given for a duration of 40 to 48 weeks and consists of BDQ, LNZ, Isoniazid (high dose), LVX, ethambutol, pyrazinamide and CFZ. Should a patient have resistance to the fluoroquinolones and/or the injectable, the patient is started on a strengthened regimen that may include BDQ, LNZ and DLM with other added agents depending on prior exposure and any other available resistance testing.

In addition to the shorter RR-TB regimen recommended by the WHO, there are other shorter regimens currently being evaluated in clinical trials. Many of these regimens employ new or re-purposed medicines such as BDQ, DLM, and LNZ, which have each been shown to be effective in clinical trials. Some of the regimens forgo the use of a second-line injectable, which is associated with a high rate of adverse events and is programmatically difficult to administer. Although these regimens are currently undergoing testing in clinical trials, the programmatic use of these regimens under operational and pragmatic research conditions can also provide important data to the global TB community about their effectiveness and safety, while also providing more information about programmatic implementation and expanding access to their potential benefits.

For this reason, BEAT Tuberculosis aims to be as pragmatic as possible, with broad eligibility criteria including almost all participants diagnosed with RR-TB. It aligns itself with the SANTP's goal to investigate an effective treatment regimen for RR-TB, while strictly adhering to the high standards of ethical conduct in clinical research. The primary objective of the trial is to evaluate the efficacy and safety of the Study Strategy, specifically to demonstrate that the intervention or Study Strategy has non-inferior efficacy to the Control Strategy.

The principle behind the Study Strategy is to "hit early and to hit hard" with the agents most likely to be effective- it is common that upon the diagnosis of RR-TB, fluoroquinolone resistance is unknown. Therefore, the Study Strategy contains three novel agents as core drugs -BDQ, LNZ, and DLM against which there is no expected Mtb resistance in the community. In addition, there are two other support medications- LVX and CFZ. Treatment will be changed on receipt of the second-line line probe assay (LPA) results. The Study Strategy has been designed to cover all possible eventualities from rifampicin mono resistant TB to Extensively Drug Resistant (XDR-TB) with an all oral regimen. The Study Strategy is given for 24 weeks but if culture conversion has not occurred by week 16, the full treatment duration can be extended to 36 weeks.

Participants include children from 6 years of age and adults diagnosed with RR-TB with or without resistance to isoniazid (INH) and/or fluoroquinolones. A total of 400 participants will be enrolled into the clinical trial. Participants will be randomized in a 1:1 ratio to receive either the Study Strategy or Control Strategy, with a stratification by clinical site and HIV status. All participants will be followed up for 76 weeks from randomization.

All patients in South Africa who are diagnosed with RR-TB are managed by the SANTP. All study tests will therefore be performed by the National Health Laboratory Services, including mycobacteriology, blood screening and safety testing and point of contact testing. These tests will be done in line with the national programme's schedule of events.

The trial will be open label, as blinding is not feasible. It is not possible to formulate placebos with multiple drugs and durations of treatment. However, the trial will be treated as if it were a blinded trial in all ways other than the physician and the participant having knowledge of the treatment assignment. Individuals assessing x-rays, cultures, ECGs and other participant information will be blinded to treatment assignment.

BEAT Tuberculosis will be conducted in Port Elizabeth in the Eastern Cape, and in Durban, KwaZulu Natal, where there is a high burden of drug resistant TB (DR TB). The clinical trial sites are established DR-TB initiation and treating sites and have been approved by the national, provincial and district TB program with the capacity for long term follow up for safety evaluation. This trial will strengthen the drug resistant TB research capacity in an under-researched area such as the Eastern Cape.

All participants will be offered an HIV test, as is standard in South Africa, and must be willing to take antiretroviral treatment, should they test positive. Wherever possible, participants who are co-infected with HIV will be managed in a joint treatment clinic to ensure close co-ordination of management of the two conditions, and to ensure that appropriate decisions can be made concerning the management of drug interactions and side effects.

Additionally, there is a pharmacokinetics/pharmacodynamics (PK-PD) aspect to the trial. There are limited data describing the association of drug concentrations with efficacy and treatment related toxicities of many of the anti-TB drugs used in the treatment of RR-TB. Understanding these PK-PD relationships can result in dose optimization to improve outcomes in the relevant patient populations. BEAT Tuberculosis is a unique opportunity to explore these relationships.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent to be enrolled in the research study prior to any study related procedures (signed or witnessed consent if the participant is unable to read and understand the informed consent document; signed or witnessed consent from a child's biological parent, legal guardian or primary caregiver) and if the participant is a child (6-17 years) is willing to sign assent
* Willing and able to adhere to the complete follow-up schedule and to study procedures
* Male or female, aged 6 years or older, including breastfeeding and/or pregnant women
* Weigh more than or equal to 16kg
* Participants above the age of 12 years, must have confirmed pulmonary TB with initial laboratory result of resistance to at least rifampicin as confirmed by genotypic or phenotypic susceptibility testing in the last three months
* Willing to use effective contraception for females of childbearing potential if sexually active; must be willing to use either an intrauterine contraceptive device or a hormonal method for the duration of the treatment regimen and for three months thereafter
* Willing to have an HIV test, and if positive, is willing to be treated with appropriate antiretroviral therapy
* Participants between the ages of 6 - 12 years, must have either confirmed pulmonary RR-TB or probable pulmonary RR-TB and a decision has been made by the referring clinician or investigator to treat the child for RR-TB
* Participants who are pregnant, should have an ultrasound done to confirm a viable intrauterine pregnancy prior to enrolment

Exclusion Criteria:

* Had taken more than 28 days but less than 24 weeks of second line TB drugs including BDQ, LNZ, CFZ, fluoroquinolones or DLM.

Please note: Participants with prior successfully treated episodes of DR TB are permitted to enroll.

* Has complicated or severe extra-pulmonary manifestations of TB, including osteo-articular, pericardial and central nervous system infection as per investigators opinion
* Is unable to take oral medication
* Is taking any prohibited medications as referred to in the protocol
* Has a known allergy or hypersensitivity to any of the medicines in the regimens
* Is currently taking part in another clinical trial of any medicinal product
* Has a QTcF interval of greater than 480 ms. Please note: If the QTcF interval is greater than 480 ms, it may be repeated if participant has reversible contributory factors, i.e. low potassium or to allow washout of previous QT prolonging drugs.
* Has clinically significant ECG abnormality in the opinion of the site investigator within 60 days prior to entry, including but not limited to second or third degree atrioventricular (AV) block or clinically important arrhythmia
* Participants with the following laboratory abnormality at screening.

  1. Haemoglobin level of < 8.0 g/dL
  2. Platelet count < 75,000/mm^3
  3. Absolute neutrophil count (ANC) < 1000/ mm^3
  4. An estimated creatinine clearance (CrCl) less than 30 mL/min as calculated by the National Health Laboratory Service (NHLS) equation
  5. Alanine aminotransferase (ALT) ≥3 x upper limit of normal (ULN)
  6. Total bilirubin grade 3 or greater (>2.0 x ULN, or >1.50 x ULN when accompanied by any increase in other liver function test)
  7. Serum potassium less than 3.2 mmol/l
* Peripheral neuropathy of grade 3 or 4 using the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events
* If in the investigator's opinion, the participant is unable to commit to study related procedures or it is unsafe for the participant to take part in the study

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2019-08-22 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
The proportion of participants with a successful outcome at the end of treatment | From 24 weeks to 76 weeks depending on assigned strategy and type of TB
  A successful treatment outcome measured at the end of treatment is defined as either Cured or Treatment Completed.
  Cured: Adequate treatment adherence (at least 80% of doses taken) as per protocol without evidence of failure and the last two negative sputum specimens at the end of treatment being culture negative. These specimens must be separated by at least 14 days.
  Treatment completed: Adequate treatment adherence (at least 80% of doses taken) as per protocol without evidence of failure but no record that two or more consecutive cultures taken at least 14 days apart are negative.
The proportion of participants with a successful outcome at the end of follow up at 76 weeks post treatment initiation | At the end of follow up at 76 weeks post treatment initiation
  A successful end of follow up outcome measured at 76 weeks post treatment initiation is defined as either Cured or Culture negative when last seen.
  Cured: Sputum Culture negative at the end of follow up at 76 weeks post treatment initiation.
  Culture negative when last seen: if the participant is lost before the end of follow up at 76 weeks and provided they have a successful treatment outcome at the last study visit attended.
The proportion of participants who experience grade 3 or greater adverse events during treatment and up to 30 days following the end of treatment | From treatment initiation to 30 days following the end of treatment
  Adverse events are graded using the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events

SECONDARY OUTCOMES:
The proportion of participants with a successful composite outcome at 76 weeks post treatment initiation | At the end of follow up at 76 weeks post treatment initiation
  A successful composite outcome is defined as a successful end of follow up outcome at 76 weeks post treatment initiation and no grade 3 or higher adverse events during treatment. A successful end of follow up outcome is either Cured or Culture negative when last seen.
PK/PD model of clofazimine exposure | Week 4
  To link PK/PD measure of Maximum Plasma Concentration (Cmax) to time to culture conversion (efficacy ) clofazimine
PK/PD model of clofazimine exposure | Week 4
  To link PK/PD measure of Area Under the Plasma Concentration-time to the time to sputum culture (efficacy) conversion for clofazimine
PK/PD model of clofazimine exposure | Week 4
  To link PK/PD measure of Concentration-time Curve From the Time of Dose Administration up to 24 Hours (AUCtime-h) to the time to sputum culture (efficacy ) conversion for clofazimine
PK/PD model of clofazimine exposure | Week 4
  To link PK/PD measure of Elimination Half-life (t1/2) to the time to sputum culture (efficacy ) conversion for clofazimine
PK/PD model of bedaquiline, delamanid, levofloxacin and linezolid exposure | Weeks 4, 12, and 24
  To link PK/PD measure of Maximum Plasma Concentration (Cmax), to culture conversion(efficacy) for bedaquiline, delamanid, levofloxacin, linezolid
PK/PD model of bedaquiline, delamanid, levofloxacin and linezolid exposure | Weeks 4, 12, and 24
  To link PK/PD measure of Time to Reach Minimum Plasma Concentration (Cmin) to the time to sputum culture (efficacy) conversion for bedaquiline, delamanid, levofloxacin, linezolid
PK/PD model of bedaquiline, delamanid, levofloxacin and linezolid exposure | Weeks 4, 12, and 24
  To link PK/PD measure of Area Under the Plasma Concentration-time Curve From the Time of Dose Administration up to 24 Hours (AUCtime-h) to the time to sputum culture (efficacy) conversion for bedaquiline, delamanid, levofloxacin, linezolid
PK/PD model of bedaquiline, delamanid, levofloxacin and linezolid exposure | Weeks 4, 12, and 24
  To link PK/PD measure of the Elimination Half-life (t1/2) to the time to sputum culture (efficacy) conversion for bedaquiline, delamanid, levofloxacin, linezolid
PK/PD model drug exposures of drugs/metabolites known to cause QT prolongation (clofazimine, bedaquiline M2 metabolite, delamanid DM6705 metabolite, and levofloxacin) | Weeks 4, 12, and 24
  To link PK/PD measure of Maximum Plasma Concentration (Cmax) to the time to toxicity of increased QTcF prolongation for clofazimine, bedaquiline M2 metabolite, delamanid DM6705 metabolite, and levofloxacin
PK/PD model drug exposures of drugs/metabolites known to cause QT prolongation (clofazimine, bedaquiline M2 metabolite, delamanid DM6705 metabolite, and levofloxacin) | Weeks 4, 12, and 24
  To link PK/PD measure of Time to Reach Maximum Plasma Concentration (Tmax),increased QTcF for clofazimine, bedaquiline M2 metabolite, delamanid DM6705 metabolite, and levofloxacin
PK/PD model drug exposures of drugs/metabolites known to cause QT prolongation (clofazimine, bedaquiline M2 metabolite, delamanid DM6705 metabolite, and levofloxacin) | Weeks 4, 12, and 24
  To link PK/PD measure of Minimum Plasma Concentration (Cmin) to the time to toxicity of increased QTcF for clofazimine, bedaquiline M2 metabolite, delamanid DM6705 metabolite, and levofloxacin
PK/PD model drug exposures of drugs/metabolites known to cause QT prolongation (clofazimine, bedaquiline M2 metabolite, delamanid DM6705 metabolite, and levofloxacin) | Weeks 4, 12, and 24
  To link PK/PD measure of the Area Under the Plasma Concentration-time Curve From the Time of Dose Administration up to 24 Hours (AUCtime-h) to the time to toxicity of increased QTcF conversion for clofazimine, bedaquiline M2 metabolite, delamanid DM6705 metabolite, and levofloxacin
PK/PD model drug exposures of linezolid | Weeks 4, 12, and 24
  To link PK/PD measures of Maximum Plasma Concentration (Cmax) to the time to toxicity of bone marrow toxicity and neuropathy
PK/PD model drug exposures of linezolid | Weeks 4, 12, and 24
  To link PK/PD measure of Time to Reach Maximum Plasma Concentration (Tmax) to the time to toxicity of bone marrow toxicity and neuropathy
PK/PD model drug exposures of linezolid | Weeks 4, 12, and 24
  To link PK/PD measure of Plasma Concentration (Cmin) to the time to toxicity of bone marrow toxicity and neuropathy
PK/PD model drug exposures of linezolid | Weeks 4, 12, and 24
  To link PK/PD measure of the Area Under the Plasma Concentration-time Curve From the Time of Dose Administration up to 24 Hours (AUCtime-h) to the time to toxicity of bone marrow toxicity and neuropathy

CONTACTS AND LOCATIONS:
Overall Officials: Francesca M Conradie, Principal Investigator — Clinical HIV Research Unit t/a Wits Health Consortium
Locations (2):
- South Africa (2):
  - Jose Pearson TB Hospital, Port Elizabeth, Eastern Cape
  - King DinuZulu Hospital Complex, Durban, KwaZulu-Natal

IPD SHARING:
Plan to Share IPD: Yes
We plan to share the de-identified individual participant data set to national and international policy makers, including the World Health Organization.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: August 2019 - August 2030
Access Criteria: There will be controlled access to the data/documents with the gatekeepers being the Principal Investigator (PI) and the chair of the Trial Steering Committee (TSC), who will be responsible for deciding who may have access. Access to the data/documents must include prior ethical approval for secondary data analysis and the statistical methods for secondary data analysis must be vetted by a statistician. If access is requested during the conduct of the trial, it must be directed to all the members of the TSC via the chair.

REFERENCES:
- [Background] Diacon AH, Pym A, Grobusch MP, de los Rios JM, Gotuzzo E, Vasilyeva I, Leimane V, Andries K, Bakare N, De Marez T, Haxaire-Theeuwes M, Lounis N, Meyvisch P, De Paepe E, van Heeswijk RP, Dannemann B; TMC207-C208 Study Group. Multidrug-resistant tuberculosis and culture conversion with bedaquiline. N Engl J Med. 2014 Aug 21;371(8):723-32. doi: 10.1056/NEJMoa1313865. PMID 25140958
- [Background] Schnippel K, Ndjeka N, Maartens G, Meintjes G, Master I, Ismail N, Hughes J, Ferreira H, Padanilam X, Romero R, Te Riele J, Conradie F. Effect of bedaquiline on mortality in South African patients with drug-resistant tuberculosis: a retrospective cohort study. Lancet Respir Med. 2018 Sep;6(9):699-706. doi: 10.1016/S2213-2600(18)30235-2. Epub 2018 Jul 11. PMID 30001994
- [Background] Sotgiu G, Centis R, D'Ambrosio L, Alffenaar JW, Anger HA, Caminero JA, Castiglia P, De Lorenzo S, Ferrara G, Koh WJ, Schecter GF, Shim TS, Singla R, Skrahina A, Spanevello A, Udwadia ZF, Villar M, Zampogna E, Zellweger JP, Zumla A, Migliori GB. Efficacy, safety and tolerability of linezolid containing regimens in treating MDR-TB and XDR-TB: systematic review and meta-analysis. Eur Respir J. 2012 Dec;40(6):1430-42. doi: 10.1183/09031936.00022912. Epub 2012 Apr 10. PMID 22496332
- [Background] Pym AS, Diacon AH, Tang SJ, Conradie F, Danilovits M, Chuchottaworn C, Vasilyeva I, Andries K, Bakare N, De Marez T, Haxaire-Theeuwes M, Lounis N, Meyvisch P, Van Baelen B, van Heeswijk RP, Dannemann B; TMC207-C209 Study Group. Bedaquiline in the treatment of multidrug- and extensively drug-resistant tuberculosis. Eur Respir J. 2016 Feb;47(2):564-74. doi: 10.1183/13993003.00724-2015. Epub 2015 Dec 2. PMID 26647431
- [Background] Drusano GL, Neely M, Van Guilder M, Schumitzky A, Brown D, Fikes S, Peloquin C, Louie A. Analysis of combination drug therapy to develop regimens with shortened duration of treatment for tuberculosis. PLoS One. 2014 Jul 8;9(7):e101311. doi: 10.1371/journal.pone.0101311. eCollection 2014. PMID 25003557
- [Background] Cox H, Ford N. Linezolid for the treatment of complicated drug-resistant tuberculosis: a systematic review and meta-analysis. Int J Tuberc Lung Dis. 2012 Apr;16(4):447-54. doi: 10.5588/ijtld.11.0451. PMID 22325685
- [Background] Briasoulis A, Agarwal V, Pierce WJ. QT prolongation and torsade de pointes induced by fluoroquinolones: infrequent side effects from commonly used medications. Cardiology. 2011;120(2):103-10. doi: 10.1159/000334441. Epub 2011 Dec 13. PMID 22156660
- [Background] Noel GJ, Goodman DB, Chien S, Solanki B, Padmanabhan M, Natarajan J. Measuring the effects of supratherapeutic doses of levofloxacin on healthy volunteers using four methods of QT correction and periodic and continuous ECG recordings. J Clin Pharmacol. 2004 May;44(5):464-73. doi: 10.1177/0091270004264643. PMID 15102866
- [Background] Diacon AH, Dawson R, von Groote-Bidlingmaier F, Symons G, Venter A, Donald PR, van Niekerk C, Everitt D, Hutchings J, Burger DA, Schall R, Mendel CM. Bactericidal activity of pyrazinamide and clofazimine alone and in combinations with pretomanid and bedaquiline. Am J Respir Crit Care Med. 2015 Apr 15;191(8):943-53. doi: 10.1164/rccm.201410-1801OC. PMID 25622149
- [Background] Denti P, Garcia-Prats AJ, Draper HR, Wiesner L, Winckler J, Thee S, Dooley KE, Savic RM, McIlleron HM, Schaaf HS, Hesseling AC. Levofloxacin Population Pharmacokinetics in South African Children Treated for Multidrug-Resistant Tuberculosis. Antimicrob Agents Chemother. 2018 Jan 25;62(2):e01521-17. doi: 10.1128/AAC.01521-17. Print 2018 Feb. PMID 29133560
- [Background] Svensson EM, Dosne AG, Karlsson MO. Population Pharmacokinetics of Bedaquiline and Metabolite M2 in Patients With Drug-Resistant Tuberculosis: The Effect of Time-Varying Weight and Albumin. CPT Pharmacometrics Syst Pharmacol. 2016 Dec;5(12):682-691. doi: 10.1002/psp4.12147. Epub 2016 Nov 8. PMID 27863179
- [Background] Svensson EM, Karlsson MO. Modelling of mycobacterial load reveals bedaquiline's exposure-response relationship in patients with drug-resistant TB. J Antimicrob Chemother. 2017 Dec 1;72(12):3398-3405. doi: 10.1093/jac/dkx317. PMID 28961790
- [Background] Gumbo T, Pasipanodya JG, Wash P, Burger A, McIlleron H. Redefining multidrug-resistant tuberculosis based on clinical response to combination therapy. Antimicrob Agents Chemother. 2014 Oct;58(10):6111-5. doi: 10.1128/AAC.03549-14. Epub 2014 Aug 4. PMID 25092691
- [Background] Chigutsa E, Pasipanodya JG, Visser ME, van Helden PD, Smith PJ, Sirgel FA, Gumbo T, McIlleron H. Impact of nonlinear interactions of pharmacokinetics and MICs on sputum bacillary kill rates as a marker of sterilizing effect in tuberculosis. Antimicrob Agents Chemother. 2015 Jan;59(1):38-45. doi: 10.1128/AAC.03931-14. Epub 2014 Oct 13. PMID 25313213
- See also: U.S. Food and Drug Administration. SIRTURO Prescribing Information — http://www.accessdata.fda.gov/drugsatfda_docs/label/2012/204384s000lbl.pdf
- See also: Bedaquiline- and delamanid- containing regimens achieve excellent interim treatment response without safety concerns — http://www.endtb.org/resources/endtb-interim-analysis-july2018
- See also: Deltyba package insert — https://www.ema.europa.eu/en/documents/product-information/deltyba-epar-product-information_en.pdf